CLINICAL TRIAL: NCT02629835
Title: A Randomized Comparison Between Intravenous and Perineural Dexamethasone for Ultrasound-Guided Axillary Blocks
Brief Title: Intravenous and Perineural Dexamethasone for Ultrasound-Guided Axillary Blocks
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montreal General Hospital (Other)
Responsible Party: Principal Investigator, De QH Tran, Associate Profesor, Montreal General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MontrealGH
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Brachial Plexus Block Duration
MeSH Terms: interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous dexamethasone 8 mg (Active Comparator): patients receiving intravenous 8 mg of dexamethasone in parallel to ultrasound guided axillary nerve block with a standardized local anesthetic solution
  Interventions: Other: intravenous 8 mg dexamethasone and perineural 0.8 ml of saline solution
- Perineural dexamethasone 8 mg (Active Comparator): patient receiving perineural 8 mg of dexamethasone in a mixture with a standardized local anesthetic solution for ultrasound guided axillary block
  Interventions: Other: intravenous 0,8 ml of saline solution and perineural 8 mg of dexamethasone

INTERVENTIONS:
Other: intravenous 8 mg dexamethasone and perineural 0.8 ml of saline solution
  Arms: Intravenous dexamethasone 8 mg
Other: intravenous 0,8 ml of saline solution and perineural 8 mg of dexamethasone
  Arms: Perineural dexamethasone 8 mg

SUMMARY:
Dexamethasone prolong the duration of brachial plexus blocks, but the optimal route, intravenous (IV) or perineural (PN), remains controversial.

This Multi-centric trial compare IV and PN dexamethasone for ultrasound-guided axillary brachial plexus blocks (AXBs). Research hypothesis is that PN modality will outlast its IV counterpart. Since analgesic duration and sensory duration can be influenced by intake of pain medications and surgical trauma to small cutaneous nerves, the investigators will select motor block duration as the main outcome.

DETAILED DESCRIPTION:
After Ethics Committee of the McGill University Health Centre, a total of 150 patients undergoing upper extremity surgery (below the elbow) will be recruited.

All AXBs will be supervised by one of the coauthors and conducted preoperatively in an induction room. This area will have full access to an oxygen source, resuscitative equipment and drugs.

All patients will have fasted for at least eight hours. An IV cannula will be placed prior the block and will be monitored and given oxygen at 2-4 L/min through nasal cannulas.

Light sedation will be provided for patient comfort if needed.Patients will be placed supine with the shoulder abducted and the elbow flexed. The AXB will have a puncture site superior to the axillary artery. After skin disinfection and draping, a skin wheal will be raised with 3 mL of lidocaine 1.5%.

In both groups, 30 mL of lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL will be used. A 22-gauge, 5 cm block will be advanced under direct US vision toward the musculocutaneous nerve. Six mL of LA will be deposited in this location. The needle will then be directed posterior to the artery, at 6 o'clock position and twenty-four mL of LA will be deposited to obtain a spread around the artery.

Patients will be randomized to receive 8 mg of IV or PN dexamethasone. In the IV group, patients will receive 0.8 mL of dexamethasone (10 mg/mL) intravenously and 0.8 mL of normal saline will be added to the injectate through the block needle. In the PN group, patients will receive 0.8 mL of normal saline intravenously and 0.8 mL of dexamethasone (10 mg/mL) will be added to the injectate through the block needle.

A research assistant will prepare the IV and PN injectates. The operator, patient and investigator assessing the block will be blinded to group allocation.

If placement of the needle tip in the desired location is unsuccessful after 15 minutes, the procedure will be stopped and the patient excluded from the study. Brachial plexus blockade will be carried out using an alternative method. If the alternative method fails as well, the patient will be given general anesthesia and intravenous narcotics will be used for postoperative analgesia

ELIGIBILITY:
Inclusion Criteria:

* Below Elbow surgery
* Age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 18 and 35 kg/m2

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or partial prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs)
* Pregnancy
* Prior surgery in the axillary region
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Motor block duration | 24 hours
  Duration of the motor block (defined as the temporal interval between the end of LA injection through the block needle and the return of movement to the hand and fingers). Patient is contacted at the next day of the surgery and asked about the time when the motor block started to disappear.

SECONDARY OUTCOMES:
duration of the sensory block | 24 hours
  defined as the temporal interval between the end of LA injection through the block needle and the return of sensation to the hand and fingers
Analgesia duration | 24 hours
  defined as the temporal interval between the end of LA injection through the block needle and the appearance of pain at the surgical site
Onset time | 30 minutes
  Time required to reach a minimal score of 14 points of a total of 16. Sensory blockade will be graded according to a 3-point scale using a cold test: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot fee touch). The cold test will be applied with light touch to avoid confusion with deep pressure sensation.
  Motor blockade will also be graded on a 3-point scale: 0 = no block, 1 = paresis, 2 = paralysis (19). Motor blockade of the musculocutaneous, radial, median and ulnar nerves will be evaluated by elbow flexion (musculocutaneous), thumb abduction (radial), thumb opposition (median) and thumb adduction (ulnar).
Success rate | 30-60 minutes
  Ability to proceed with surgery without the need for intravenous narcotics, general anesthesia, rescue blocks or LA infiltration by the surgeon. Just propofol based sedation (25-80 μg/kg/min) will be permitted if necessary, keeping always response to verbal stimulus.

OTHER OUTCOMES:
Demographic data | 30 minutes
  sex, age, weight, height, type of surgery
Side effects | 30-60 minutes
  vascular puncture, hematoma at the site of puncture, toxic effects of LA
Persistent deficit | 7 days
  All patients will be contacted after 7 days by a blinded observer asking about persistent sensory or motor deficit in relation with the blocked nerves.

CONTACTS AND LOCATIONS:
Overall Officials: De QH Tran, MD, FRCPC, Principal Investigator — Associate Professor
Locations (3):
- Montreal General Hospital, McGill University, Montreal, Quebec, Canada
- Thailand (2):
  - Ramathibodi Hospital, Mahidol University,, Bangkok, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Chiang Mai

REFERENCES:
- [Background] Persec J, Persec Z, Kopljar M, Zupcic M, Sakic L, Zrinjscak IK, Marinic DK. Low-dose dexamethasone with levobupivacaine improves analgesia after supraclavicular brachial plexus blockade. Int Orthop. 2014 Jan;38(1):101-5. doi: 10.1007/s00264-013-2094-z. Epub 2013 Sep 6. PMID 24173676
- [Result] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Result] Tandoc MN, Fan L, Kolesnikov S, Kruglov A, Nader ND. Adjuvant dexamethasone with bupivacaine prolongs the duration of interscalene block: a prospective randomized trial. J Anesth. 2011 Oct;25(5):704-9. doi: 10.1007/s00540-011-1180-x. Epub 2011 Jun 17. PMID 21681533
- [Result] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Result] Kawanishi R, Yamamoto K, Tobetto Y, Nomura K, Kato M, Go R, Tsutsumi YM, Tanaka K, Takeda Y. Perineural but not systemic low-dose dexamethasone prolongs the duration of interscalene block with ropivacaine: a prospective randomized trial. Local Reg Anesth. 2014 Apr 5;7:5-9. doi: 10.2147/LRA.S59158. eCollection 2014. PMID 24817819
- [Result] Shrestha BR, Maharjan SK, Tabedar S. Supraclavicular brachial plexus block with and without dexamethasone - a comparative study. Kathmandu Univ Med J (KUMJ). 2003 Jul-Sep;1(3):158-60. PMID 16388222
- [Result] Yadav RK, Sah BP, Kumar P, Singh SN. Effectiveness of addition of neostigmine or dexamethasone to local anaesthetic in providing perioperative analgesia for brachial plexus block: A prospective, randomized, double blinded, controlled study. Kathmandu Univ Med J (KUMJ). 2008 Jul-Sep;6(23):302-9. doi: 10.3126/kumj.v6i3.1704. PMID 20071811
- [Result] Parrington SJ, O'Donnell D, Chan VW, Brown-Shreves D, Subramanyam R, Qu M, Brull R. Dexamethasone added to mepivacaine prolongs the duration of analgesia after supraclavicular brachial plexus blockade. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):422-6. doi: 10.1097/AAP.0b013e3181e85eb9. PMID 20814282
- [Result] Biradar PA, Kaimar P, Gopalakrishna K. Effect of dexamethasone added to lidocaine in supraclavicular brachial plexus block: A prospective, randomised, double-blind study. Indian J Anaesth. 2013 Mar;57(2):180-4. doi: 10.4103/0019-5049.111850. PMID 23825819
- [Result] Abdallah FW, Johnson J, Chan V, Murgatroyd H, Ghafari M, Ami N, Jin R, Brull R. Intravenous dexamethasone and perineural dexamethasone similarly prolong the duration of analgesia after supraclavicular brachial plexus block: a randomized, triple-arm, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):125-32. doi: 10.1097/AAP.0000000000000210. PMID 25629321
- [Result] Movafegh A, Razazian M, Hajimaohamadi F, Meysamie A. Dexamethasone added to lidocaine prolongs axillary brachial plexus blockade. Anesth Analg. 2006 Jan;102(1):263-7. doi: 10.1213/01.ane.0000189055.06729.0a. PMID 16368840
- [Result] Yaghoobi S, Seddighi M, Yazdi Z, Ghafouri R, Khezri MB. Comparison of Postoperative Analgesic Effect of Dexamethasone and Fentanyl Added to Lidocaine through Axillary Block in Forearm Fracture. Pain Res Treat. 2013;2013:761583. doi: 10.1155/2013/761583. Epub 2013 Dec 29. PMID 24490067
- [Result] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Result] Tran DQ, Bertini P, Zaouter C, Munoz L, Finlayson RJ. A prospective, randomized comparison between single- and double-injection ultrasound-guided infraclavicular brachial plexus block. Reg Anesth Pain Med. 2010 Jan-Feb;35(1):16-21. doi: 10.1097/AAP.0b013e3181c7717c. PMID 20048654
- [Result] Gonzalez AP, Bernucci F, Pham K, Correa JA, Finlayson RJ, Tran DQ. Minimum effective volume of lidocaine for double-injection ultrasound-guided axillary block. Reg Anesth Pain Med. 2013 Jan-Feb;38(1):16-20. doi: 10.1097/AAP.0b013e3182707176. PMID 23146999
- [Derived] Aliste J, Leurcharusmee P, Engsusophon P, Gordon A, Michelagnoli G, Sriparkdee C, Tiyaprasertkul W, Tran DQ, Van Zundert TC, Finlayson RJ, Tran DQH. A randomized comparison between intravenous and perineural dexamethasone for ultrasound-guided axillary block. Can J Anaesth. 2017 Jan;64(1):29-36. doi: 10.1007/s12630-016-0741-8. Epub 2016 Sep 23. PMID 27663451